CLINICAL TRIAL: NCT02380846
Title: The Metabolic Effects of Consuming Carbohydrate With Different Protein Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2013/00589
Record Dates: First submitted 2015-01-28; First posted 2015-03-05 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases | interventions — In Situ Hybridization, Fluorescence; Egg White

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Rice (Other): Control session - white rice (equivalent to 50g available carbohydrates)
  Interventions: Other: White rice
- Rice with chicken (Active Comparator): Treatment 1 - White rice and steamed chicken breast (25g protein)
  Interventions: Other: Rice with chicken breast
- Rice with fish (Active Comparator): Treatment 2 - White rice and steamed fish (25g protein)
  Interventions: Other: Rice with fish
- Rice with egg white (Active Comparator): Treatment 3 - White rice and egg white (25g protein)
  Interventions: Other: Rice with egg white
- Rice with beancurd (Active Comparator): Treatment 4 - White rice and steamed beancurd (25g protein)
  Interventions: Other: Rice with beancurd

INTERVENTIONS:
Other: White rice — Control - white rice
  Arms: Rice
Other: Rice with chicken breast — Treatment 1 - steamed white rice with steamed chicken breast
  Arms: Rice with chicken
Other: Rice with fish — Treatment 2 - steamed white rice with steamed fish
  Arms: Rice with fish
Other: Rice with egg white — Treatment 3 - steamed white rice with egg white
  Arms: Rice with egg white
Other: Rice with beancurd — Treatment 4 - steamed white rice with steamed beancurd
  Arms: Rice with beancurd

SUMMARY:
This study aims to find out how consuming different proteins with rice affect metabolism. Most meals the investigators eat predominantly consist of a carbohydrate and protein (i.e. rice, noodles, bread etc with meats or seafood). However, it is still unknown how consuming different proteins with commonly eaten carbohydrates affect metabolism. Previous studies have shown that proteins stimulate hormones such as insulin, glucagon and gut hormones. However, the extent of the response depends on protein type. The metabolic responses to carbohydrates have also been shown to be greatly affected when they are eaten with proteins. However, most of the previous studies have used glucose as the carbohydrate and it is still unknown how eating proteins with carbohydrate foods such as rice affect metabolism. Therefore, this study has been initiated to determine the metabolic effects of eating different protein types with rice. Using the most common carbohydrate eaten in Asia (rice) and four commonly eaten protein foods (egg, chicken, fish and beancurd), this study aims to observe the metabolic effects of co-ingesting proteins and carbohydrate. The resulting data will provide valuable insights into the metabolic effects of protein-carbohydrate meals and will be useful in the development of practical advice and dietary guidelines for those with chronic diseases (such as diabetes and obesity).

DETAILED DESCRIPTION:
The study will recruit 20 healthy Chinese male subjects from the general public over a period of one year. The test foods will be rice, rice with egg, rice with fish, rice with chicken and rice with beancurd.Potential participants will have to come on one morning in an overnight fasted state for consenting and screening procedures. Only those fulfilling the inclusion and exclusion criteria will be admitted into the study. Each participant will be required to come on 5 non-consecutive days, with each session lasting approximately 4 hours. On each day, participants will arrive at the laboratory between 8-9 am following an overnight fast. An indwelling catheter will be inserted into a vein in their forearm or antecubital fossa and kept patent. Baseline blood samples will be obtained after which they will be given the test food to consume. Further blood samples will be taken at periodic intervals for the subsequent 3.5 hours. Blood samples will be taken every 15 minutes in the first 60 minutes and every 30 minutes for the remaining 150 minutes. At every time point blood samples will be extracted from a finger prick (for measuring glucose) and from the cannula (for measuring all other metabolites). At the same time points subjects will have to fill in visual analogue scales on feelings of hunger and satiety.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Male
* Age between 21-40 years
* Do not have any metabolic diseases (diabetes, hypertension etc)
* Do not have G6PD deficiency
* Not on prescription medication known to affect glucose related metabolism
* Not allergic/intolerant to any of the test foods
* Do not partake in sports at the competitive and/or endurance levels
* Weight of at least 45kg
* Body mass index between 18.0 to 24.9 kg/m2
* Normal blood pressure (120/80 mmHg)
* Fasting blood glucose <6.0 mmol/L

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Blood glucose response (incremental area under the curve) measured using the hemocue | 3.5 hours post consumption
  Blood glucose response (incremental area under the curve) measured using the hemocue
Insulin (incremental area under the curve) is determined using the COBAS | 3.5 hours post consumption
  Insulin (incremental area under the curve) is determined using the COBAS
Glucagon determined using the ELISA | 3.5 hours post consumption
  Glucagon is determined using the ELISA

SECONDARY OUTCOMES:
Effects of physical activity | Assessed at the start of every test session 1-2 weekly and up to 8 weeks in total per subject.
  Self-reported evaluation of physical activity according to a qualitative scale: light, medium or strenuous exercise done the day before the study visit.
Satiety: Hunger and fullness measured using the Visual analogue scale | Assessed at the start of every test session 1-2 weekly and up to 8 weeks in total per subject.
  Hunger and fullness measured using the Visual Analogue Scale